CLINICAL TRIAL: NCT02753062
Title: Multicenter Phase II Study of Bendamustine Plus Subcutaneous Rituximab in Patients With Diffuse Large B-cell Lymphoma (DLBCL) Type Monomorphic Post-transplant Lymphoproliferative Disorder
Brief Title: Bendamustine Plus Subcutaneous Rituximab in Patients With Diffuse Large B-cell Lymphoma
Acronym: PTLD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Cheolwon Suh (Unknown)
Responsible Party: Principal Investigator, Dok Hyun Yoon, Assistant professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR_PTLD
Record Dates: First submitted 2016-04-08; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bendamustine, rituximab (Experimental): Bendamustine plus subcutaneous Rituximab treatment of 6 cycles. Rituximab 1400mg subcutaneous over 5mins on day 1 and bendamustine 120mg/m2 + NS 500mL iv over 1hour on day 1 and 2.
  Interventions: Drug: bendamustine, rituximab

INTERVENTIONS:
Drug: bendamustine, rituximab — subjects will receive rituximab 375mg/m2 on day 1 and bendamustine 120mg/m2 by intravenous infusion on day 2 and 3 in the first cycle. From the 2nd to 6th cycle, rituximab will be administered subcutaneously at a fixed dose of 1400mg and bendamustine 120mg/m2 by intravenous infusion on day 1 following administration of rituximab and day 2.
  Other Names: symbenda, mabthera

SUMMARY:
This is an open-label, multi-center, prospective, single arm phase 2 trial of the combination of bendamustine and rituximab in patients with PTLD, monomorphic cluster of differentiation antigen 20(CD20) positive DLBCL. The investigators want to investigate the efficacy and safety of the combination of bendamustine and rituximab in patients with previously untreated PTLD, monomorphic CD20 (+) diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Monomorphic PTLD comprise more than 70% of PTLDs and diffuse large B-cell lymphoma is the predominant subtype. However, none of the trials have been performed for the specific population of DLBCL type monomorphic PTLD. The investigators will select Patients with proven, measurable monomorphic PTLD of DLBCL after solid organ transplantation (e.g. heart, lung, liver or kidney etc.). Patients having PTLD with or without Epstein-Barr virus (EBV) association, positive for CD20 monomorphic DLBCL type. The B-R treatment will continue up to 6 cycles with interval of 21 days. Patients will receive 375 mg/m2 on day 1 and bendamustine 120 mg/m2 by intravenous infusion on day 2 and 3 in the first cycle. From the 2nd to 6th cycle, rituximab will be administered subcutaneously at a fixed dose of 1400 mg and bendamustine 120 mg/m2 by intravenous infusion on day 1 following administration of rituximab and day 2. On the first day of infusion of bendamustine in each cycle, palonosetron 0.25 mg will be given as a single intravenous injection about 30 minutes before infusion of bendamustine. Pegfilgrastim 6 mg will be administered as a single subcutaneous injection between 24 to 48 hours after completion of chemotherapy at each cycle. Based on relatively good safety profile and efficacy of bendamustine and rituximab (BR regimen), the investigators will investigate a feasibility of BR regimen in this immunocompromised patients with DLBCL type monomorphic PTLD.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Histologically confirmed adult patients diagnosed with CD20-positive monomorphic PTLD, DLBCL irrespective of EBV association
3. Patients having undergone solid organ transplantation (heart, lung, liver, kidney, pancreas, small intestine transplantation, etc or a combination of the organ transplantations mentioned).
4. No prior treatment for PTLD, DLBCL except reduction of immunosuppression
5. At least one measurable lesion ≥ 1.5 cm in greatest transverse diameter by spiral CT
6. Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2.
7. Age ≥ 19
8. Adequate renal function: serum creatinine level < 2.0 mg/dL
9. Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value (or < 5 x ULN in the presence of DLBCL involvement of the liver), bilirubin < 2 X upper normal value (or < 5 x ULN in the presence of DLBCL involvement of the liver)
10. Adequate hematological function: hemoglobin ≥ 9.0 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL, unless abnormalities are due to bone marrow involvement by lymphoma. (Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment).
11. Life expectancy 6 months
12. A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are < 1 years after the onset of menopause.
13. Female patients of child bearing potential must use an effective method of birth control (i.e. hormonal contraceptive, intrauterine device,diaphragm with spermicide, condom with spermicide or abstinence) during treatment period and 12 month thereafter; Males must use an effective method of birth control during treatment period and 12 months thereafter.

Exclusion Criteria:

1. Other subtypes PTLD than monomorphic CD20 (+) DLBCL
2. Previous treatment for PTLD, DLBCL with immunotherapy or chemotherapy except for short-term corticosteroids (duration of ≤ 8 days) before inclusion (Low dose steroid as immunosuppressant are allowed.)
3. central nervous system (CNS) involvement by lymphoma or any evidence of spinal cord compression.
4. Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin, early gastric cancer or carcinoma in situ of the cervix or breast or untreated prostatic cancer without any plan for a treatment) unless the patient has been free of the disease for ≥ 3 years
5. Patients with a known history of HIV or HCV seropositivity.
6. Patients with active hepatitis B i. HBsAg positive or ii. HBsAg negative, anti-HBc-Ab positive and HBV-DNA PCR positive patients
7. Pregnant or lactating women
8. Men who are not surgically sterile or women of childbearing potential not employing adequate contraception
9. Other serious illness or medical conditions i. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months ii. History of significant neurological or psychiatric disorders including dementia or seizures iii. Active, uncontrolled infections requiring systemic antibiotic therapy or other serious infections within 14 days before study enrollment iv. Other serious medical illnesses
10. Known hypersensitivity to any of the study drugs or its ingredients
11. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 6 to 8 weeks after completion of the 6th cycle of treatment.

SECONDARY OUTCOMES:
Assess response rate | 2 to 3 weeks (or start of next cycle) after completion of the 3rd cycle of treatment and 6 to 8 weeks after completion of the 6th cycle of treatment.
Assess event-free survival | the time from the 1st day of treatment to the first recording of disease-progression, relapse or death of any cause or failure to achieve CR after completion, assessed up to 96 months
Assess overall survival | the time from the 1st day of treatment to death of any cause or the date of last follow-up, assessed up to 96 months.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From the date of first drug administration until the date of the 28th days of last drug administration, assessed up to 22 weeks
Assess health-related quality of life by EORTC QLQ-C30 (3rd edition) | within 14 days prior to treatment start and every 12 months (± 1 months) of follow-up period until final analysis and at the time of disease progression, assessed up to 96 months

CONTACTS AND LOCATIONS:
Overall Officials: Wonseog Kim, M.D., PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
we will share collected data with principal investigators in Korea